CLINICAL TRIAL: NCT05598632
Title: Risk Factors for Stroke or Systemic Embolism in Chinese Patients with Non-Valvular Atrial Fibrillation Registry
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-CXGC09-1
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Stroke; Atrial fibrillation; Risk factors; Registry
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is aimed to validate the existing stroke risk stratification model for patients with atrial fibrillation (AF) (CHA2DS2-VASc Score, CHADS2 Score, ATRIA score, ABC score, etc.) and establish a new stroke risk assessment model using a nationwide AF -specific registry in China.

DETAILED DESCRIPTION:
This study is a multicenter prospective disease-specific registry of patients with atrial fibrillation (AF) that will analyze factors that are associated with stroke or systemic embolic events in patients with AF in China. Approximately 5,000 prospective cohort of patients and 22,000 retrospective cohort of patients will be enrolled. Consecutive patients who meet the eligibility criteria and provide informed consent. Patients enrolled in the registry will be followed for approximately 3 years. Patient follow-up by National Center for Cardiovascular Diseases will continue as scheduled. Atrial Fibrillation Data capture will include demographics, cardiovascular risk factors, diagnosis, type of AF (paroxysmal, persistent, permanent AF), treatment strategy (rate vs. rhythm), antithrombotic therapy, concomitant medications and doses, laboratory tests, echo and computed tomography results, blood sample, insurance and provider information, comorbidities, and outcomes. The primary outcome will be stroke or non-CNS embolism. Other pre-defined outcomes of interest will include major adverse cardiac events, all-cause mortality, cause-specific death (sudden, non-sudden, heart failure-related), major bleeding, and hospitalization for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older; male or female.
* History of documented atrial fibrillation.
* Able to provide written informed consent.

Exclusion Criteria:

* Subjects with moderate or severe mitral stenosis or a mechanical heart valve
* Subjects with previous or planned AF ablation.
* Subjects with previous or planned left atrial appendage closure.
* Subjects unable to cooperate with follow-up after assessment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients without valvular heart disease, prevous/planned ablation or left atrial appendage closure.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Stroke and Systemic Embolic Events (SEE) | At 12-month after recruiting
  The composite of stroke and Systemic Embolic Events (SEE) during follow-up. A stroke is defined as an abrupt onset, over minutes to hours, of a focal neurologic deficit that is generally in the distribution of a single brain artery (including the retinal artery) and that is not due to an identifiable nonvascular cause (ie, brain tumor or trauma).
  A systemic embolic event is defined as an abrupt episode of arterial insufficiency associated with clinical or radiologic evidence of arterial occlusion in the absence of other likely mechanisms (eg, atherosclerosis, instrumentation). Arterial embolic events involving the central nervous system (including the eye), coronary, and pulmonary arterial circulation are not considered SEEs,. Diagnosis of embolism to the lower extremities requires arteriographic demonstration of abrupt arterial occlusion.

SECONDARY OUTCOMES:
Major Bleeding Events | At 12-month after recruiting
  A major bleeding event is defined as clinically overt bleeding event (ie, bleeding that is visualized by examination or radiologic imaging) that meets ≥1 of the following:
  1. Fatal bleeding
  2. Symptomatic bleeding in a critical area or organ such as:
     * Retroperitoneal
     * Intracranial
     * Intraocular
     * Intraspinal
     * Intraarticular
     * Pericardial
     * Intramuscular with compartment syndrome
All-Cause Mortality | At 12-month after recruiting
  All-Cause Mortality during follow-up
Cardiac Death | At 12-month after recruiting
  Cardiac Death during follow-up
Hospitalization for heart failure | At 12-month after recruiting
  Hospitalization for heart failure during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD, PhD, Study Chair — Fuwai Hospital, Chinese Academy of Medical Science
Locations (1):
- Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Qi W, Yuan S, Liu H, Xu M, Yang Y, Peng X, Hu Z, Zhang Y, Zhao Y, Zheng L, Yao Y, Zheng Z; Investigators the REFINE Registry; investors. Rationale, design and protocol for risk factors for stroke in patients with non-valvular atrial fibrillation in China: a nationwide registry (REFINE registry). BMJ Open. 2025 Nov 4;15(11):e104806. doi: 10.1136/bmjopen-2025-104806. PMID 41193204